CLINICAL TRIAL: NCT01247376
Title: Temperature Sensitive Release of PGE2 and Diminished Energy Requirements in Synovial Tissue With Postoperative Cryotherapy - A Prospective Randomised Study After Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Dr Anders Stålman
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2007/59-31/4
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Knee Arthroscopy; Meniscus; Inflammation; Hydrops; Cooling
Keywords: inflammation; arthroscopy; knee; microdialysis
MeSH Terms: conditions — Inflammation; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Cooling and compression (No Intervention)
- Intervention with cooling and compression (Experimental)
  Interventions: Device: Cooling and compression

INTERVENTIONS:
Device: Cooling and compression — Cooling and compression of the knee postoperatively with an Aircast device.
  Arms: Intervention with cooling and compression

SUMMARY:
Abstract

Background:

Local external cooling of the postoperative field is a treatment paradigm aiming for enhanced recovery after joint surgery. It is supposed to reduce pain and improve mobilization, enabling same day surgery.

Hypothesis:

Systematic postoperative cooling and compression after knee arthroscopy will reduce pain and also be reflected by changes in local levels of metabolic and inflammatory variables in the synovial membrane.

Study design:

Prospective randomised study; Level of evidence 1.

Methods:

Forty-four otherwise healthy patients were included in the study and randomised to systematic cooling and compression or NO cooling and compression after knee arthroscopy. Microdialysis of the synovial membrane was performed postoperatively with measurements of PGE2, glucose, lactate, glycerol, glutamate and blood flow (ethanol exchange ratio). Local temperature was monitored as well as postoperative pain (VAS and NRS).

Results:

The application of a cooling and compression device after knee arthroscopy resulted in significantly lower temperature in the operated knee (skin, joint capsule and intraarticularly).

The cooling and compression diminished energy requirements in synovial tissue and a 3 temperature sensitive influence on inflammation (PGE2) were shown. No effect on postoperative pain was detected.

Conclusion:

Local cryotherapy and compression after knee arthroscopy significantly lowered local knee temperature postoperatively. A correlation with synovial PGE 2 and temperature was shown.

Since PGE2 is a pain and inflammatory marker this implicates a positive anti-inflammatory effect induced by postoperative local cooling and compression. Hypothermia is proposed to have a protective effect in ischemic tissue. This is probably due to a decreased metabolic rate and therefore decreased energy requirements as shown by stable levels of lactate despite lower blood flow indicated by increasing ethanol ratio.

ELIGIBILITY:
Inclusion Criteria:

* indication for knee arthroscopy due to suspected meniscus injury

Exclusion Criteria:

* osteoarthritis or known systemic inflammatory disease, eg RA

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Synovial measurements of metabolic and inflammatory markers (glucose, lactate, glutamate, PGE2)

SECONDARY OUTCOMES:
Subjective pain measurements (Visual analogue scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden, Sweden

REFERENCES:
- [Background] Raynor MC, Pietrobon R, Guller U, Higgins LD. Cryotherapy after ACL reconstruction: a meta-analysis. J Knee Surg. 2005 Apr;18(2):123-9. doi: 10.1055/s-0030-1248169. PMID 15915833
- [Background] Stalman A, Tsai JA, Segerdahl M, Dungner E, Arner P, Fellander-Tsai L. Ketorolac but not morphine exerts inflammatory and metabolic effects in synovial membrane after knee arthroscopy: a double-blind randomized prospective study using the microdialysis technique. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):557-64. doi: 10.1097/aap.0b013e3181bfbd9f. PMID 19916211
- [Background] Stalman A, Tsai JA, Wredmark T, Dungner E, Arner P, Fellander-Tsai L. Local inflammatory and metabolic response in the knee synovium after arthroscopy or arthroscopic anterior cruciate ligament reconstruction. Arthroscopy. 2008 May;24(5):579-84. doi: 10.1016/j.arthro.2007.12.010. Epub 2008 Feb 20. PMID 18442691
- [Background] Fellander-Tsai L, Hogberg E, Wredmark T, Arner P. In vivo physiological changes in the synovial membrane of the knee during reperfusion after arthroscopy. A study using the microdialysis technique. J Bone Joint Surg Br. 2002 Nov;84(8):1194-8. doi: 10.1302/0301-620x.84b8.13187. PMID 12463670